CLINICAL TRIAL: NCT00851760
Title: Idiopathic Epiretinal Macular Membrane and Cataract Extraction : Combined vs Consecutive Surgery
Brief Title: Epiretinal Macular Membrane and Cataract Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Pr Creuzot Garcher, Centre Hospitalier Universitaire Dijon
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU Dijon OPH 01
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: Epiretinal Macular Membrane; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Combined Surgery (Experimental)
  Interventions: Procedure: Combined surgery
- 2 consecutive surgery (Active Comparator)
  Interventions: Procedure: Consecutive surgery

INTERVENTIONS:
Procedure: Consecutive surgery — Consecutive surgery for epiretinal macular membrane and cataract extraction
  Arms: 2 consecutive surgery
Procedure: Combined surgery — Combined surgery for epiretinal macular membrane and cataract extraction
  Arms: 1 Combined Surgery

SUMMARY:
The investigators proposed to assess the functional and anatomical outcomes of cataract and idiopathic epiretinal macular membrane extraction in combined and consecutive surgeries.

DETAILED DESCRIPTION:
A retrospective nonrandomized clinical case series study collected 174 consecutive eyes of 174 patients undergoing macular surgery between January 2005 and December 2006. Patients suffering from epiretinal macular membranes (ERM) secondary to uveitis, trauma, or associated with a simultaneous retinal detachment (RD) were excluded. We treated 109 eyes with a combined procedure (group 1) and 65 eyes with a consecutive surgery (membrane surgery and cataract separately)(group 2).

ELIGIBILITY:
Inclusion Criteria:

* All patients had symptomatic visual loss and needed vitrectomy for ERM removal.

Exclusion Criteria:

* Patients suffering from ERM secondary to uveitis, trauma, or associated with a simultaneous RD were excluded.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Combined and consecutive surgeries are effective procedures to treat idiopathic ERM. The functional and anatomical results are equivalent in both procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmology Unit CHU Dijon, Dijon, Burgundy, France